CLINICAL TRIAL: NCT02357979
Title: Fissure Caries Inhibition Study With Solea CO2-9.3μm Short-pulsed Laser - A Randomized, Single Blind, Prospective, Split Mouth Controlled, Clinical Trial
Brief Title: Fissure Caries Inhibition Study With Solea CO2-9.3μm Short-pulsed Laser
Acronym: LaserFissure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LaserFissure-1st
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Dental Caries
Keywords: caries; prevention; laser; fluoride
MeSH Terms: conditions — Dental Caries | interventions — Lasers; Fluorides

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Laser & Fluoride (Experimental): In the split mouth design the molar on one side of the mouth receives the intervention CO2 9.3 μm short pulsed laser treatment and fluoride varnish (experimental side) in the occlusal fissure areas.
  Interventions: Device: Laser
- Fluoride alone (Active Comparator): In the split mouth design this arm (this side in the mouth - the contralateral tooth to the experimental site in the same jaw) will receive only fluoride varnish treatment. In the split mouth design this opposite side of the jaw is functioning as control.
  Interventions: Other: Fluoride

INTERVENTIONS:
Device: Laser — CO2 - 9.3μm short-pulsed laser irradiation will occur on the occlusal enamel surface. This results in changes in crystal composition and structure, which increase the resistance of dental mineral to dissolution by acid and will work to better prevent dental caries in the occlusal surface of vital teeth when compared to fluoride therapy alone over 12 months.
  Other Names: Convergent Solea CO2 laser
  Arms: Laser & Fluoride
Other: Fluoride — The Fluoride varnish is painted on the occlusal surface of the tooth. Fluoride varnish makes enamel more acid resistant.
  Arms: Fluoride alone

SUMMARY:
The objective of this clinical study is to evaluate whether the use of the new CO2 - 9.3μm short-pulsed laser increases the caries resistance of occlusal pit and fissure surfaces in patients in addition to fluoride therapy. This will be quantified by visual exams with the International Caries Detection and Assessment System (ICDAS II), SOPROLIFE daylight and blue fluorescence, and DIAGNOdent Laser Light-induced Fluorescence. This is a randomized, single blind, prospective, split mouth controlled, clinical trial over 12 months.

DETAILED DESCRIPTION:
The study is designed as randomized, single blind, prospective, split mouth controlled, clinical trial over 12 months. The subjects for this study will be recruited from the UCSF School of Dentistry. Patients meeting the inclusion criteria from the UCSF Predoctoral, Postgraduate Pediatric Dental and Postgraduate orthodontic clinics will have the study explained to them and be invited to participate.

Young patients with moderate/high caries risk will be invited to enroll into the study. They will have to have a pair of two molars which have not been treated so far and are caries free and not sealed. The molar on patient's dominant side (right or left) will be randomly assigned to either the test or the control group with the contralateral non-dominant side receiving the other treatment. The test tooth will be treated with CO2 laser irradiation and fluoride varnish; the control tooth will receive fluoride varnish treatment alone.

A baseline visual inspection using ICDAS II, white and blue light digital photographs (SOPROLIFE), and DIAGNOdent assessments will be made by a dentist prior to treatment.

The patient will be asked to return for a 6-month and a 12-month follow up exam, at which time visual inspection with all testing methods will be conducted by the dentist who originally completed the baseline exam. The endpoint of the study for each participant will be when either the control or test tooth is found to have significant demineralization by ICDAS assessment (ICDAS code 3 - "localized enamel breakdown without clinical visual signs of dentinal involvement") or at the 12 month exam, whichever comes first.

The control and test teeth might be sealed with a dental sealant at the end of the study. All data obtained will be analyzed for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* age 6 or older, in good general health
* subject is of moderate or high caries risk according to CAMBRA
* has at least one pair of unsealed molars in at least one jaw with need for a sealant
* teeth with an ICDAS code 0, 1 and 2 with deep grooves and fissures providing an anatomical stick for an explorer
* willing to comply with all study procedures and protocols
* must be able to read and understand English
* have an understanding of the study
* residing in San Francisco or other nearby locales with community water fluoridation (to eliminate water fluoridation as a potential confounding variable)
* patient and parent/guardian able to provide written informed consent in English
* willing to sign the "Authorization for Release of Personal Health Information and Use of Personally Unidentified Study Data for Research" form; data will only be used for research.

Exclusion Criteria:

* show evidence of extremely poor oral hygiene
* subjects suffering from systemic diseases, significant past or medical history with conditions that may affect oral health or oral flora (i.e. diabetes, HIV, heart conditions that require antibiotic prophylaxis),
* taking medications that may affect the oral flora or salivary flow (e.g. antibiotic use in the past three months, drugs associated with dry mouth / xerostomia [extreme high caries risk])
* other conditions that may decrease the likelihood of adhering to study protocol
* subjects who will leave the area and are unable to complete the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rechmann, DDS, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF School of Dentistry - Dental Offices in Bay Area, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Beltran-Aguilar ED, Barker LK, Canto MT, Dye BA, Gooch BF, Griffin SO, Hyman J, Jaramillo F, Kingman A, Nowjack-Raymer R, Selwitz RH, Wu T; Centers for Disease Control and Prevention (CDC). Surveillance for dental caries, dental sealants, tooth retention, edentulism, and enamel fluorosis--United States, 1988-1994 and 1999-2002. MMWR Surveill Summ. 2005 Aug 26;54(3):1-43. PMID 16121123
- [Background] Brown LJ, Kaste LM, Selwitz RH, Furman LJ. Dental caries and sealant usage in U.S. children, 1988-1991: selected findings from the Third National Health and Nutrition Examination Survey. J Am Dent Assoc. 1996 Mar;127(3):335-43. doi: 10.14219/jada.archive.1996.0203. PMID 8819780
- [Background] Lussi A. Validity of diagnostic and treatment decisions of fissure caries. Caries Res. 1991;25(4):296-303. doi: 10.1159/000261380. PMID 1913769
- [Background] Featherstone JD. Caries detection and prevention with laser energy. Dent Clin North Am. 2000 Oct;44(4):955-69, ix. PMID 11048282
- [Background] Pitts NB. How the detection, assessment, diagnosis and monitoring of caries integrate with personalized caries management. Monogr Oral Sci. 2009;21:1-14. doi: 10.1159/000224208. Epub 2009 Jun 3. PMID 19494672
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] de Josselin de Jong E, Sundstrom F, Westerling H, Tranaeus S, ten Bosch JJ, Angmar-Mansson B. A new method for in vivo quantification of changes in initial enamel caries with laser fluorescence. Caries Res. 1995;29(1):2-7. doi: 10.1159/000262032. PMID 7867045
- [Background] Al-Khateeb S, Forsberg CM, de Josselin de Jong E, Angmar-Mansson B. A longitudinal laser fluorescence study of white spot lesions in orthodontic patients. Am J Orthod Dentofacial Orthop. 1998 Jun;113(6):595-602. doi: 10.1016/s0889-5406(98)70218-5. PMID 9637561
- [Background] Tranaeus S, Al-Khateeb S, Bjorkman S, Twetman S, Angmar-Mansson B. Application of quantitative light-induced fluorescence to monitor incipient lesions in caries-active children. A comparative study of remineralisation by fluoride varnish and professional cleaning. Eur J Oral Sci. 2001 Apr;109(2):71-5. doi: 10.1034/j.1600-0722.2001.00997.x. PMID 11347658
- [Background] Tranaeus S, Shi XQ, Lindgren LE, Trollsas K, Angmar-Mansson B. In vivo repeatability and reproducibility of the quantitative light-induced fluorescence method. Caries Res. 2002 Jan-Feb;36(1):3-9. doi: 10.1159/000057583. PMID 11961323
- [Background] Pretty IA, Ellwood RP. Comparison of paired visual assessment and software analyses of changes in caries status over 6 months from fluorescence images. Caries Res. 2007;41(2):115-20. doi: 10.1159/000098044. PMID 17284912
- [Background] Yin W, Feng Y, Hu D, Ellwood RP, Pretty IA. Reliability of quantitative laser fluorescence analysis of smooth surface lesions adjacent to the gingival tissues. Caries Res. 2007;41(3):186-9. doi: 10.1159/000099316. PMID 17426397
- [Background] Rocha RO, Ardenghi TM, Oliveira LB, Rodrigues CR, Ciamponi AL. In vivo effectiveness of laser fluorescence compared to visual inspection and radiography for the detection of occlusal caries in primary teeth. Caries Res. 2003 Nov-Dec;37(6):437-41. doi: 10.1159/000073396. PMID 14571122
- [Background] Astvaldsdottir A, Holbrook WP, Tranaeus S. Consistency of DIAGNOdent instruments for clinical assessment of fissure caries. Acta Odontol Scand. 2004 Aug;62(4):193-8. doi: 10.1080/00016350410001612. PMID 15513415
- [Background] Tranaeus S, Lindgren LE, Karlsson L, Angmar-Mansson B. In vivo validity and reliability of IR fluorescence measurements for caries detection and quantification. Swed Dent J. 2004;28(4):173-82. PMID 15779494
- [Background] Bamzahim M, Aljehani A, Shi XQ. Clinical performance of DIAGnodent in the detection of secondary carious lesions. Acta Odontol Scand. 2005 Feb;63(1):26-30. doi: 10.1080/00016350510019621. PMID 16095059
- [Background] Angnes V, Angnes G, Batisttella M, Grande RH, Loguercio AD, Reis A. Clinical effectiveness of laser fluorescence, visual inspection and radiography in the detection of occlusal caries. Caries Res. 2005 Nov-Dec;39(6):490-5. doi: 10.1159/000088185. PMID 16251794
- [Background] Reis A, Mendes FM, Angnes V, Angnes G, Grande RH, Loguercio AD. Performance of methods of occlusal caries detection in permanent teeth under clinical and laboratory conditions. J Dent. 2006 Feb;34(2):89-96. doi: 10.1016/j.jdent.2005.04.002. Epub 2005 Jun 20. PMID 15970371
- [Background] Akarsu S, Koprulu H. In vivo comparison of the efficacy of DIAGNOdent by visual inspection and radiographic diagnostic techniques in the diagnosis of occlusal caries. J Clin Dent. 2006;17(3):53-8. PMID 17022365
- [Background] Rechmann P, Rechmann BM, Featherstone JD. Caries detection using light-based diagnostic tools. Compend Contin Educ Dent. 2012 Sep;33(8):582-4, 586, 588-93; quiz 594, 596. PMID 22953601
- [Background] Rechmann P, Charland D, Rechmann BM, Featherstone JD. Performance of laser fluorescence devices and visual examination for the detection of occlusal caries in permanent molars. J Biomed Opt. 2012 Mar;17(3):036006. doi: 10.1117/1.JBO.17.3.036006. PMID 22502564
- [Background] Hafstrom-Bjorkman U, Sundstrom F, de Josselin de Jong E, Oliveby A, Angmar-Mansson B. Comparison of laser fluorescence and longitudinal microradiography for quantitative assessment of in vitro enamel caries. Caries Res. 1992;26(4):241-7. doi: 10.1159/000261446. PMID 1423438
- [Background] Emami Z, al-Khateeb S, de Josselin de Jong E, Sundstrom F, Trollsas K, Angmar-Mansson B. Mineral loss in incipient caries lesions quantified with laser fluorescence and longitudinal microradiography. A methodologic study. Acta Odontol Scand. 1996 Feb;54(1):8-13. doi: 10.3109/00016359609003502. PMID 8669246
- [Background] al-Khateeb S, ten Cate JM, Angmar-Mansson B, de Josselin de Jong E, Sundstrom G, Exterkate RA, Oliveby A. Quantification of formation and remineralization of artificial enamel lesions with a new portable fluorescence device. Adv Dent Res. 1997 Nov;11(4):502-6. doi: 10.1177/08959374970110041801. PMID 9470510
- [Background] al-Khateeb S, Oliveby A, de Josselin de Jong E, Angmar-Mansson B. Laser fluorescence quantification of remineralisation in situ of incipient enamel lesions: influence of fluoride supplements. Caries Res. 1997;31(2):132-40. doi: 10.1159/000262388. PMID 9118185
- [Background] Ferreira Zandona AG, Analoui M, Beiswanger BB, Isaacs RL, Kafrawy AH, Eckert GJ, Stookey GK. An in vitro comparison between laser fluorescence and visual examination for detection of demineralization in occlusal pits and fissures. Caries Res. 1998;32(3):210-8. doi: 10.1159/000016455. PMID 9577987
- [Background] Lussi A, Imwinkelried S, Pitts N, Longbottom C, Reich E. Performance and reproducibility of a laser fluorescence system for detection of occlusal caries in vitro. Caries Res. 1999 Jul-Aug;33(4):261-6. doi: 10.1159/000016527. PMID 10343088
- [Background] Shi XQ, Welander U, Angmar-Mansson B. Occlusal caries detection with KaVo DIAGNOdent and radiography: an in vitro comparison. Caries Res. 2000 Mar-Apr;34(2):151-8. doi: 10.1159/000016583. PMID 10773633
- [Background] Shi XQ, Tranaeus S, Angmar-Mansson B. Validation of DIAGNOdent for quantification of smooth-surface caries: an in vitro study. Acta Odontol Scand. 2001 Apr;59(2):74-8. doi: 10.1080/000163501750157153. PMID 11370753
- [Background] Altenburger MJ, Gmeiner B, Hellwig E, Wrbas KT, Schirrmeister JF. The evaluation of fluorescence changes after application of casein phosphopeptides (CPP) and amorphous calcium phosphate (ACP) on early carious lesions. Am J Dent. 2010 Aug;23(4):188-92. PMID 21250566
- [Background] Featherstone JD, Nelson DG. Laser effects on dental hard tissues. Adv Dent Res. 1987 Oct;1(1):21-6. doi: 10.1177/08959374870010010701. No abstract available. PMID 3125842
- [Background] Kantorowitz Z, Featherstone JD, Fried D. Caries prevention by CO2 laser treatment: dependency on the number of pulses used. J Am Dent Assoc. 1998 May;129(5):585-91. doi: 10.14219/jada.archive.1998.0276. PMID 9601171
- [Background] Goodis HE, Fried D, Gansky S, Rechmann P, Featherstone JD. Pulpal safety of 9.6 microm TEA CO2 laser used for caries prevention. Lasers Surg Med. 2004;35(2):104-10. doi: 10.1002/lsm.20043. PMID 15334612
- [Background] Gorton J, Featherstone JD. In vivo inhibition of demineralization around orthodontic brackets. Am J Orthod Dentofacial Orthop. 2003 Jan;123(1):10-4. doi: 10.1067/mod.2003.47. PMID 12532056
- [Background] Rechmann P, Fried D, Le CQ, Nelson G, Rapozo-Hilo M, Rechmann BM, Featherstone JD. Caries inhibition in vital teeth using 9.6-mum CO2-laser irradiation. J Biomed Opt. 2011 Jul;16(7):071405. doi: 10.1117/1.3564908. PMID 21806251
- [Background] Rechmann P, Charland DA, Rechmann BM, Le CQ, Featherstone JD. In-vivo occlusal caries prevention by pulsed CO2 -laser and fluoride varnish treatment--a clinical pilot study. Lasers Surg Med. 2013 Jul;45(5):302-10. doi: 10.1002/lsm.22141. Epub 2013 Jun 4. PMID 23737079
- [Background] Zuerlein MJ, Fried D, Featherstone JD. Modeling the modification depth of carbon dioxide laser-treated dental enamel. Lasers Surg Med. 1999;25(4):335-47. doi: 10.1002/(sici)1096-9101(1999)25:43.0.co;2-f. PMID 10534750
- [Background] Featherstone JD, Nelson DG. Recent uses of electron microscopy in the study of physico-chemical processes affecting the reactivity of synthetic and biological apatites. Scanning Microsc. 1989 Sep;3(3):815-27; discussion 827-8. PMID 2617263
- [Background] Takagi S, Liao H, Chow LC. Effect of tooth-bound fluoride on enamel demineralization/ remineralization in vitro. Caries Res. 2000 Jul-Aug;34(4):281-8. doi: 10.1159/000016603. PMID 10867429
- [Background] Young DA, Featherstone JD. Caries management by risk assessment. Community Dent Oral Epidemiol. 2013 Feb;41(1):e53-63. doi: 10.1111/cdoe.12031. PMID 24916678
- [Background] Terrer E, Koubi S, Dionne A, Weisrock G, Sarraquigne C, Mazuir A, Tassery H. A new concept in restorative dentistry: light-induced fluorescence evaluator for diagnosis and treatment. Part 1: Diagnosis and treatment of initial occlusal caries. J Contemp Dent Pract. 2009 Nov 1;10(6):E086-94. PMID 20020086
- [Background] Terrer E, Raskin A, Koubi S, Dionne A, Weisrock G, Sarraquigne C, Mazuir A, Tassery H. A new concept in restorative dentistry: LIFEDT-light-induced fluorescence evaluator for diagnosis and treatment: part 2 - treatment of dentinal caries. J Contemp Dent Pract. 2010 Jan 1;11(1):E095-102. PMID 20098972
- [Derived] Rechmann P, Kubitz M, Chaffee BW, Rechmann BMT. Fissure caries inhibition with a CO2 9.3-mum short-pulsed laser-a randomized, single-blind, split-mouth controlled, 1-year clinical trial. Clin Oral Investig. 2021 Apr;25(4):2055-2068. doi: 10.1007/s00784-020-03515-x. Epub 2020 Aug 15. PMID 32803438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed between February 2018 and November 2019 at the University of California, San Francisco (UCSF) School of Dentistry.
Units Other Than Participants: 2nd molars-2/subject- 1-side L&F other F
Period: Overall Study
Arm/Group | Laser & Fluoride | Fluoride Alone
Started (Each participant provided two units - one right, one left second molar) | 60; 60 2nd molars-2/subject- 1-side L&F other F | 60; 60 2nd molars-2/subject- 1-side L&F other F
Completed | 55; 55 2nd molars-2/subject- 1-side L&F other F | 55; 55 2nd molars-2/subject- 1-side L&F other F
Not Completed | 5; 5 2nd molars-2/subject- 1-side L&F other F | 5; 5 2nd molars-2/subject- 1-side L&F other F
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Population: Each participant had to provide a cavity free pair of second molars (right and left second molar in one jaw (upper or lower jaw) - only ICDAS scores 0, 1 and 2 were allowed at baseline for these teeth.
Units Other Than Participants: right or left second molar
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser & Fluoride | Fluoride Alone | Total
Number analyzed (Participants) | 60 | 60 | 60
Number analyzed (right or left second molar) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 60 | 120
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (1.4) | 13.1 (1.4) | 13.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 28 | 28 | 56
Race (NIH/OMB) [Count of Units; unit: right or left second molar]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 16 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 31 | 31 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: right or left second molar]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: International Caries Detection and Assessment System (ICDAS II) - Number of Molars With ICDAS Score of 3 or More - ICDAS Score 3, Cavity -
Description: Difference in number of lesion changes into ICDAS score 3 (signifying a cavity) between matched case and control teeth (within patient) from baseline to 6 months and baseline to 12 months.
  The International Caries Detection and Assessment System (ICDAS) is a visual assessment of the caries levels. The ICDAS score ranges from 0 to 6, with score 0 meaning no demineralization at all, score 3 means a first physical loss of enamel, and score 6 means a huge cavity.
Time Frame: 1 year
Measure: Count of Units; unit: right or left second molar
Units Other Than Participants: right or left second molar
Arm/Group | Laser & Fluoride | Fluoride Alone
Number analyzed (Participants) | 55 | 55
Number analyzed (right or left second molar) | 55 | 55
right or left second molar | 0 | 13

2. Primary Outcome: Change in ICDAS Scores - International Caries Detection and Assessment System (ICDAS II) -
Description: Differences in change in ICDAS scores between matched case and control teeth (within patient) from baseline to 6 months and baseline to 12 months.
  The International Caries Detection and Assessment System (ICDAS) is a visual assessment of the caries levels. The ICDAS score ranges from 0 to 6, with the score 0 meaning no demineralization at all, score 3 means a first physical loss of enamel, and score 6 means a huge cavity.
Time Frame: 1 year
Measure: Count of Units; unit: right or left molar
Units Other Than Participants: right or left molar
Arm/Group | Laser & Fluoride | Fluoride Alone
Number analyzed (Participants) | 51 | 51
Number analyzed (right or left molar) | 51 | 51
right or left molar
  ICDAS score change -1 | 4 | 0
  ICDAS score change 0 | 34 | 13
  ICDAS score change +1 | 12 | 28
  ICDAS score change +2 | 1 | 10

3. Secondary Outcome: Change in SOPROlife Scores
Description: Differences in change in SOPROlife scores between matched case and control teeth (within patient) from baseline to 6 months and baseline to 12 month.
  The SOPROlife score (name of the intraoral camera system) is a visual assessment of the caries levels. The SOPROlife score ranges from 0 to 6, with score 0 meaning no demineralization at all, and score 6 means a huge cavity.
Time Frame: 1 year
Measure: Count of Units; unit: right or left second molar
Units Other Than Participants: right or left second molar
Arm/Group | Laser & Fluoride | Fluoride Alone
Number analyzed (Participants) | 52 | 51
Number analyzed (right or left second molar) | 52 | 51
right or left second molar
  change -1 | 2 | 0
  change 0 | 47 | 19
  change +1 | 1 | 30
  change +2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment through one year follow up.
Arm/Group | Laser & Fluoride | Fluoride Alone
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT02357979/Prot_SAP_000.pdf